CLINICAL TRIAL: NCT00287963
Title: A Phase I Study of Topotecan in Combination With Vinorelbine in Recurrent Lung Cancer
Brief Title: Topotecan and Vinorelbine in Treating Patients With Recurrent Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454919; MUSC-104864/725; GSK-100780
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; combined type small cell lung cancer; intermediate type small cell lung cancer; large cell lung cancer; lymphocyte-like type small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Topotecan; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinorelbine + topotecan (Experimental)
  Interventions: Drug: topotecan hydrochloride; Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: topotecan hydrochloride
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan and vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of topotecan when given together with vinorelbine in treating patients with recurrent lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of topotecan when combined with vinorelbine ditartrate in patients with recurrent lung cancer.

Secondary

* Assess the response and stable disease rates and the time to disease progression among treated patients.

OUTLINE: This is a dose-escalation study of topotecan.

Patents receive vinorelbine ditartrate IV over 8-10 minutes and topotecan IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which ≥ 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed lung cancer

  * All histologic types eligible
  * Recurrent or progressive disease after ≥ 1 prior chemotherapy regimen with or without radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) ≤ 2
* Karnofsky PS ≥ 60%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other active invasive malignancy
* No uncontrolled illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No psychiatric illness/social situation that would limit compliance with study requirements
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to topotecan or vinorelbine ditartrate

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy
* No prior therapy with topotecan or vinorelbine ditartrate
* No chemotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* Recovered from agents administered > 4 weeks earlier
* No other concurrent investigational agents
* No concurrent palliative radiotherapy
* No other concurrent anticancer therapies or agents
* No concurrent hormones or other chemotherapy except for the following:

  * Steroids for adrenal failure
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)
  * Intermittent dexamethasone as an antiemetic

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Cycle 1 (up to day 21)

SECONDARY OUTCOMES:
Response rate | while on study, at the end of each 3 week cycle
stable disease rate | while on study, at the end of each 3 week cycle
time to progression | from start of treatment to day of documented progression or death, whichever comes first, up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Study Chair — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Beldner MA, Sherman CA, Green MR, Garrett-Mayer E, Chaudhary U, Meyer ML, Kraft AS, Montero AJ. Phase I dose escalation study of vinorelbine and topotecan combination chemotherapy in patients with recurrent lung cancer. BMC Cancer. 2007 Dec 20;7:231. doi: 10.1186/1471-2407-7-231. PMID 18096059